CLINICAL TRIAL: NCT03827213
Title: Prospective Randomized Control Trial Evaluating Single Shot Exparel Versus Indwelling Interscalene Catheter for Total Shoulder Replacements- A Pilot Study
Brief Title: Exparel Interscalene vs Indwelling Catheter
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ran out of medication
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Elilary Montilla Medrano, Assistant Professor of Anesthesiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-9707
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Pain
Keywords: shoulder surgery, post operative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single shot Interscalene Nerve Block (Experimental): This group will receive an interscalene nerve block. This will be administered as a single 20mL injection consisting of a mixture of 10mL of Exparel and 10mL of 0.5% bupivacaine hydrochloride.
  Interventions: Drug: Exparel
- Indwelling Interscalene Catheter (Active Comparator): This group will receive an indwelling interscalene catheter placed posterior to C5-C6 nerve roots (between the shoulders) and administered 15 mL of 0.5% ropivacaine plain for the block with no superficial cervical block. The "On-Q" pump will be set at a rate of 4 mL/hr.
  Interventions: Device: Indwelling Interscalene Catheter

INTERVENTIONS:
Drug: Exparel — A shot of long acting local anesthetic for post operative pain management
  Other Names: liposomal bupivacaine
  Arms: Single shot Interscalene Nerve Block
Device: Indwelling Interscalene Catheter — ropivacaine, given through a catheter inserted between the shoulders
  Arms: Indwelling Interscalene Catheter

SUMMARY:
The investigators are comparing an indwelling catheter with intermediate duration local anesthetic to a single shot peripheral nerve block with long acting a local anesthetic (Exparel).

DETAILED DESCRIPTION:
While placing an indwelling nerve catheter can prolong pain control, it can also have drawbacks and complications. While major complications like pneumothorax and hemidiaphragmatic paresis from interscalene continuous peripheral nerve blocks (CPNB) are rare, minor adverse effects associated with CPNBs may be more common. They include infection and anatomical damage to blood vessels and nerves due to the indwelling catheter. In addition, catheters take a significantly longer time to set up and place than single shot blocks, which is important as there is often a rush to block patients and trying to get them into the operating room on time. Furthermore, the needle used for catheter placement is larger than the single shot needles, which creates more discomfort to patients during the nerve block. The catheter itself is taped around the entire sides and back of the patient's neck, which is also uncomfortable for patients. Because of how shallow the interscalene block is, the catheter is often found to be dislodged from operating room positioning, patient transport or movement, which negates the placement of the catheter. An indwelling catheter must also be followed up by the acute pain service team until the catheter is removed.

Exparel, or liposomal bupivacaine, is formulated to release low dose bupivacaine over 96 hours, and was recently approved by the FDA in April 2018 to be used in interscalene blocks. The sustained release of local anesthetic could theoretically act similarly to the continuous infusion of local anesthetic through an indwelling interscalene catheter, and could thus avoid the need for placement of a catheter. Current existing data, although inconclusive, has in some studies shown an equal analgesic effect as catheters. As per pharmacy, the cost of the On-Q pump and the local anesthesia needed for the pump together cost $390 for each indwelling catheter placed, not including the cost of anesthesia and pharmacy supplies and labor. The cost of each 20 mL vial of Exparel is less at $285 and, for a single shot nerve block, would avoid the extra costs and time needed for a catheter placement.

The investigators would like to perform a prospective randomized controlled pilot study to examine the efficacy of single shot interscalene blocks using Exparel versus the traditional interscalene catheter used at our institution. The purpose of the study the investigators are proposing is to determine if single shot interscalene nerve blocks using Exparel can provide equivalent or better analgesia than indwelling interscalene catheter in patients who undergo total shoulder replacement surgery. If so, single shot interscalene nerve blocks with Exparel may serve as a quicker, easier, cheaper, safer, and more comfortable alternative to placing indwelling interscalene catheters.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) 1, 2, and 3
* Ages 40-74
* Patients scheduled for total shoulder replacement

Exclusion Criteria:

* ASA 4 and 5
* Pre-existing pain disorder
* Regular consumption of chronic pain medication
* pregnant women
* any medical condition such as a clotting disorder
* anatomic abnormality that precludes use of an indwelling scalene catheter
* Body Mass Index (BMI) >40
* Patient refusal
* Pre-existing diabetic neuropathy or Hemoglobin A1c >9
* Failed block

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elilary Montilla Medrano, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borgeat A, Ekatodramis G. Anaesthesia for shoulder surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):211-25. doi: 10.1053/bean.2002.0234. PMID 12491553
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Wiegel M, Gottschaldt U, Hennebach R, Hirschberg T, Reske A. Complications and adverse effects associated with continuous peripheral nerve blocks in orthopedic patients. Anesth Analg. 2007 Jun;104(6):1578-82, table of contents. doi: 10.1213/01.ane.0000261260.69083.f3. PMID 17513661
- [Background] Sabesan VJ, Shahriar R, Petersen-Fitts GR, Whaley JD, Bou-Akl T, Sweet M, Milia M. A prospective randomized controlled trial to identify the optimal postoperative pain management in shoulder arthroplasty: liposomal bupivacaine versus continuous interscalene catheter. J Shoulder Elbow Surg. 2017 Oct;26(10):1810-1817. doi: 10.1016/j.jse.2017.06.044. Epub 2017 Aug 24. PMID 28844420
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Shot Interscalene Nerve Block: This group received an interscalene nerve block. This was administered as a single 20mL injection consisting of a mixture of 10mL of Exparel and 10mL of 0.5% bupivacaine hydrochloride.
- Indwelling Interscalene Catheter: This group received an indwelling interscalene catheter placed posterior to C5-C6 nerve roots (between the shoulders) and administered 15 mL of 0.5% ropivacaine plain for the block with no superficial cervical block. The "On-Q" pump was set at a rate of 4 mL/hr.
Period: Overall Study
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Started | 11 | 12
Completed | 7 | 11
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirements Assessed at 24 Hours Post-surgery
Description: Participant opioid requirements at 24 hours from treatment in morphine equivalents. Will report how much pain management medication participant needed within first 24 hours post-surgery.
Time Frame: 24 Hours post-surgery
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Intra-Operative Opioid Requirements
Description: Opioid requirements (morphine equivalents) during surgery. Will report how much pain management medication participant needed during surgery.
Time Frame: Duration of Surgery (Approximately 3 hours)
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Opioid Requirements Assessed at 8-hours Post-surgery
Description: 8-hour Opioid requirements (morphine equivalents). Will report how much pain management medication participant needed within first 8 hours after surgery.
Time Frame: 8 hour post-surgery
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Score in Post Anesthesia Care Unit (PACU)
Description: Collecting patient pain scores in the Post Anesthesia Care Unit (PACU). Participant will be asked to rate their pain score from 0 (no pain) to10 (worst pain)
Time Frame: During time in PACU (up to 5 hours)
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Opioid Requirements Assessed at 48 Hours Post-surgery
Description: 48 hour Opioid requirements (morphine equivalents). Will report how much pain management medication participant needed within first 48 hours after surgery.
Time Frame: 48 hours post-surgery
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Length of Stay
Description: Number of days subjects stayed until discharge. Will report how many days participant stayed in hospital after surgery.
Time Frame: At Discharge (up to 3 days)
Population: Data were not collected/aggregated and, as such, no data was available for analysis of Outcome Measure.
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 72 hours
Arm/Group | Single Shot Interscalene Nerve Block | Indwelling Interscalene Catheter
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Interscalene Nerve Block (N=11) | Indwelling Interscalene Catheter (N=12)
Postoperative Respiratory Complications (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Shortness of Breath
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 1 (1) | 0 (0) — Chest Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT03827213/Prot_SAP_000.pdf